CLINICAL TRIAL: NCT01112267
Title: A Randomized, Placebo-Controlled, Parallel Group, Double-Blind Clinical Study to Evaluate the Efficacy and Safety of Tramadol HCl/Acetaminophen Extended Release Tablet in Subjects With Chronic Low Back Pain
Brief Title: An Efficacy and Safety Study of Extended Release (ER) Tramadol Hydrochloride (HCl)/Acetaminophen in Participants With Chronic Low-Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR016222; ULTER-KOR-3003; TRAMAPPAI3004
Record Dates: First submitted 2010-04-01; First posted 2010-04-28 (Estimated); Results first posted 2013-07-24 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-06

CONDITIONS: Low Back Pain
Keywords: Chronic low back pain; Tramadol Hydrochloride (HCl); acetaminophen
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tramadol Hydrochloride (HCl)/acetaminophen (Experimental): Participants will receive 1 tablet containing fixed dose of combination of tramadol hydrochloride (HCl) 75 milligram (mg) /acetaminophen Extended Release (ER) 650 mg orally once daily on Days 1 to 3, 1 tablet twice daily (tramadol HCl 150 mg/acetaminophen 1300 mg) on Days 4 to 7, then 1 or 2 tablets twice daily on Days 8 to 28.
  Interventions: Drug: Tramadol HCl/acetaminophen Extended Release
- Placebo (Placebo Comparator): Prticipants will receive 1 tablet matching placebo once daily orally on Days 1 to 3, 1 tablet twice daily on Days 4 to 7, then 1 or 2 tablets twice daily on Days 8 to 28.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tramadol HCl/acetaminophen Extended Release — Participants will receive 1 tablet containing 75 mg of tramadol HCl and 650 mg of acetaminophen, once daily on Days 1to 3, then 1 tablet twice daily on Days 4 to 7
  Other Names: Ultracet Extended Relaese
  Arms: Tramadol Hydrochloride (HCl)/acetaminophen
Drug: Placebo — Participants will receive 1 matching placebo tablet once daily on Days 1 to 3, then 1 tablet twice daily on Days 4 to 7
  Arms: Placebo
Drug: Tramadol HCl/acetaminophen Extended Release — Participants will receive 1 or 2 tablets containing 75 mg of tramadol HCl and 650 mg of acetaminophen, twice daily on Days 8 to 28
  Other Names: Ultracet Extended Relaese
  Arms: Tramadol Hydrochloride (HCl)/acetaminophen
Drug: Placebo — Prticipants will receive 1 or 2 matching placebo tablet once daily on Days 1 to 3, then 1 tablet twice daily on Days 8 to 28
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of extended release (ER) tramadol hydrochloride (HCl)/acetaminophen compared with placebo in participants with chronic (lasting a long time) low-back pain.

DETAILED DESCRIPTION:
This is a double blind (a medical research study in which neither the researchers nor the participants know what treatment the participants is receiving), randomized (study drug is assigned by chance), placebo-controlled, parallel group (a medical research study comparing the response in 2 or more groups of participants receiving different interventions [treatments]) and up-titration study in participants with chronic low back pain. The study will consist of 6 visits (Day -7 to Day -1 [Visit 1], Day 1 [Visit 2], Day 3 [telephone visit], Day 8 [Visit 3], Day 15 [Visit 4] and Day 29 [Visit 5]) and 2 phases: a screening phase and treatment phase. Screening phase will be of 7 days during which, participants will receive stable dose of non-steroidal anti-inflammatory drugs (NSAIDS) or COX-2 selective inhibitors (NSAID that specifically inhibits an enzyme known as cyclooxygenase-2) for pain therapy. On the basis of average pain intensity over the last 48 hours which will be measured at baseline (at the end of screening period), participants will enter the treatment phase. Treatment phase will be of 28 days which includes 7-days of dose titration period. In treatment phase all participants will be randomly assigned to 1 of 2 possible treatments: tramadol HCl 75 milligram (mg)/acetaminophen 650 mg ER tablet treatment or the equivalent placebo (an inactive substance) treatment until study completion, Day 29. Participants will receive 1 tablet of tramadol HCl/acetaminophen ER or its equivalent placebo, once daily for 3 days. After the first 3 days, the participants will receive a telephone inquiry monitoring the occurrence of adverse events and will be given additional administration instructions for the next 4 days (1 tablet twice daily for 4 days). From Day 7, participants will receive 1 or 2 tablets twice a day depending on the degree of pain relief required. Participants will visit the center on the Day 8 (Visit 3), Day 15 (Visit 4), and Day 29 (Visit 5) after starting study drug. The efficacy will be assessed by measuring extent of reduction in pain intensity on a Visual Analog Scale (VAS). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with low back pain at least 3 months before the screening or washout period
* Participants who have taken a stable dose of Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) (drugs used for reducing inflammation and pain ) or Cyclo-Oxygenase 2 (COX-2) selective inhibitors (an anti-inflammatory drug that fights pain) from 7 days before investigational product administration, and could maintain the same dose during the period of the study
* Participants whose average pain intensity is more than or equal to 4.0 centimeters on Visual Analog Scale over the last 48 hours after the completion of screening
* Postmenopausal or surgically sterile or abstinent women or practicing a highly effective method of birth control
* Women with childbearing potential must have negative pregnancy test

Exclusion Criteria:

* Participants who have taken tramadol or tramadol HCl or acetaminophen, or narcotic (strong habit-forming drug that stops pain and depresses the central nervous system) analgesic tablet within 30 days before investigational product administration
* Participants who have taken acetaminophen tablet within 7 days before investigational product administration
* Participants with tumor or infection in meninges or spinal cord
* Participants who have fibromyalgia (neurosensory disorder characterized by muscle pain, joint stiffness, and fatigue), reflex sympathetic dystrophy (feeling of pain associated with evidence of minor nerve injury) or causalgia (persistent, severe burning sensation of the skin), acute spinal cord compression, acute nerve root compression, severe lower extremity weakness or numbness, regional pain syndrome, meningitis (inflammation of the meninges), diskitis (nonbacterial inflammation of an intervertebral disk or disk space), back pain because of secondary infection or tumor, or pain caused by a confirmed or suspected neoplasm
* Participants who have taken analgesic (including local agents or anesthetics), sedative-hypnotic (e.g., diazepam), or muscle relaxant other than a stable dose of NSAIDs or COX-2 selective inhibitors within 5 times the half-life of the concerned agent before investigational product administration

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.

REFERENCES:
- [Derived] Lee JH, Lee CS; Ultracet ER Study Group. A randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of the extended-release tramadol hydrochloride/acetaminophen fixed-dose combination tablet for the treatment of chronic low back pain. Clin Ther. 2013 Nov;35(11):1830-40. doi: 10.1016/j.clinthera.2013.09.017. Epub 2013 Oct 30. PMID 24183364

RESULTS

PARTICIPANT FLOW:
Groups:
- Tramadol HCl/Acetaminophen: Participants received 1 tablet containing fixed dose of combination of tramadol hydrochloride (HCl) 75 milligram (mg) /acetaminophen Extended Release (ER) 650 mg orally once daily on Days 1 to 3, 1 tablet twice daily (tramadol HCl 150 mg/acetaminophen 1300 mg) on Days 4 to 7, then 1 or 2 tablets twice daily on Days 8 to 28.
- Placebo: Participants received 1 tablet of matching placebo once daily orally on Days 1 to 3, 1 tablet twice daily on Days 4 to 7, then 1 or 2 tablets twice daily on Days 8 to 28.
Period: Overall Study
Arm/Group | Tramadol HCl/Acetaminophen | Placebo
Started | 126 | 122
Treated | 125 | 120
Completed | 92 | 104
Not Completed | 34 | 18
Not completed — Adverse Event | 24 | 6
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Protocol Violation | 5 | 3
Not completed — Participants not compliant | 1 | 2
Not completed — Participants not receive any study drug | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tramadol HCl/Acetaminophen | Placebo | Total
Number analyzed (Participants) | 125 | 120 | 245
Age Continuous [Mean (Standard Deviation); unit: Years] | 59.93 (10.72) | 60.39 (9.87) | 60.16 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 89 | 183
  Male | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Reduction in Pain Intensity
Description: The percentage of participants with extent of reduction in pain intensity greater than or equal to 30 percent was reported. Pain intensity change rate was calculated by Visual Analog Scale (VAS) score at baseline minus VAS score at Day 29 divided by VAS score at Baseline. VAS is a 10 centimeter (cm) scale. Intensity of pain range: 0 cm=no pain to 10 cm=worst possible pain.
Time Frame: Baseline up to Day 29
Population: Full analysis set (FAS) population included all participants who had received investigational product and had at least 1 data of measurement of primary efficacy endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tramadol HCl/Acetaminophen | Placebo
Number analyzed (Participants) | 85 | 90
Percentage of Participants | 57.65 [47.14 to 68.15] | 41.11 [30.95 to 51.28]
Statistical Analysis 1: Comparison: Tramadol HCl/Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.0367, Cochran-Mantel-Haenszel; p-value for percentage of participants with reduction in pain intensity was calculated for tramadol HCl/acetaminophen and placebo groups

2. Primary Outcome: Change From Baseline in Pain Intensity at Day 29
Description: Change in pain intensity experienced by participants over the last 48 hours was measured on Day 29 against Baseline with VAS. VAS is a 10 cm scale. Intensity of pain range: 0 cm=no pain to 10 cm=worst possible pain.
Time Frame: Baseline and Day 29
Population: The FAS population included all the participants who had received investigational product and had at least 1 data of measurement of primary efficacy endpoint.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Tramadol HCl/Acetaminophen | Placebo
Number analyzed (Participants) | 85 | 90
Unit on a scale
  Baseline | 6.334 (1.383) | 6.000 (1.331)
  Change at Day 29 | 2.299 (1.764) | 1.549 (1.578)
Statistical Analysis 1: Comparison: Tramadol HCl/Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.0095, Mann-Whitney U test — p-value for change in reduction in pain intensity at Day 29 was calculated for tramadol HCl/acetaminophen and placebo groups

3. Secondary Outcome: Percentage of Participants With Pain Relief
Description: Pain relief was measured in 6 stages to assess the participant's pain relief. Extent of pain relief was measured on a scale ranging from 4 to -1, where 4=complete disappearance, 3=fair relief, 2=moderate relief, 1=slight relief, 0=no change and -1=pain worsening. Relief more than 'slight relief (1)' was considered as pain relief success.
Time Frame: Day 8, Day 15 and Day 29
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tramadol HCl/Acetaminophen | Placebo
Number analyzed (Participants) | 85 | 90
Percentage of participants
  Day 8: Slight relief (n=82,88) | 70.73 [60.88 to 80.58] | 53.41 [42.99 to 63.83]
  Day 15: Slight relief (n=85,89) | 82.35 [74.25 to 90.46] | 65.17 [55.27 to 75.07]
  Day 29, Slight relief (85,89) | 81.18 [72.87 to 89.49] | 77.53 [68.86 to 86.20]
Statistical Analysis 1: Comparison: Tramadol HCl/Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.0202, Chi-squared — p-value for percentage of participants with pain relief at Day 8 was calculated for tramadol HCl/acetaminophen and placebo groups
Statistical Analysis 2: Comparison: Tramadol HCl/Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.0102, Chi-squared — p-value for percentage of participants with pain relief at Day 15 was calculated for tramadol HCl/acetaminophen and placebo groups
Statistical Analysis 3: Comparison: Tramadol HCl/Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.4652, Chi-squared — p-value for percentage of participants with pain relief at Day 29 was calculated for tramadol HCl/acetaminophen and placebo groups

4. Secondary Outcome: Change From Baseline in Short Form (SF)-36 Score at Day 29
Description: The quality of life of participants was evaluated by SF-36 Korean version questionnaire. It is composed of 8 domains: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. Participants answered to the questionnaire of 36 questions; and physical, social, and psychological health status were assessed. It ranges 0 to 100, and higher score indicates better quality of life, But in "Reported (Rptd.) Health Transition" domain higher score indicates worse quality of life.
Time Frame: Baseline and Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Tramadol HCl/Acetaminophen | Placebo
Number analyzed (Participants) | 85 | 90
Unit on a scale
  Baseline: Physical functioning | 46.71 (20.71) | 47.94 (20.80)
  Change at Day 29: Physical functioning (n=83,87) | 9.82 (18.35) | 6.67 (15.99)
  Baseline: Role physical | 44.93 (24.18) | 49.51 (26.17)
  Change at Day 29: Role Physical (n=83,87) | 16.04 (23.89) | 8.69 (22.62)
  Baseline: Bodily pain | 34.66 (14.46) | 35.99 (13.89)
  Change at Day 29: Bodily pain (n=83,87) | 19.39 (18.99) | 17.69 (14.84)
  Baseline: General health | 43.56 (17.92) | 48.11 (17.05)
  Change at Day 29: General health (n=83,87) | 7.36 (14.41) | 2.77 (12.58)
  Baseline: Vitality | 38.82 (19.93) | 42.71 (17.83)
  Change at Day 29: Vitality (n=83,87) | 11.14 (20.55) | 5.82 (18.94)
  Baseline: Social functioning | 64.26 (22.59) | 64.58 (26.98)
  Change at Day 29: Social functioning (n=83,87) | 11.75 (25.70) | 6.61 (20.60)
  Baseline: Role emotional | 61.76 (27.41) | 61.57 (29.34)
  Change at Day 29: Role emotional (n=83,87) | 8.13 (28.93) | 7.47 (28.25)
  Baseline: Mental Health | 61.06 (19.03) | 60.56 (19.34)
  Change at Day 29: Mental Health (n=83,87) | 20.48 (23.20) | 18.39 (24.61)
  Baseline: Rptd. health transition | 65.00 (24.76) | 63.61 (20.92)
  Change at Day 29: Rptd. health transition(n=83,87) | -18.07 (25.99) | -6.90 (30.19)
Statistical Analysis 1: Comparison: Tramadol HCl/Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.3524, Wilcoxon (Mann-Whitney) — p-value for change from Baseline in physical conditioning at Day 29 was calculated using for tramadol HCl/acetaminophen and placebo groups
Statistical Analysis 2: Comparison: Tramadol HCl/Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.0224, Wilcoxon (Mann-Whitney) — p-value for change from Baseline in role physical at Day 29 was calculated for tramadol HCl/acetaminophen and placebo groups
Statistical Analysis 3: Comparison: Tramadol HCl/Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.5712, Wilcoxon (Mann-Whitney) — p-value for change from Baseline in bodily pain at Day 29 was calculated for tramadol HCl/acetaminophen and placebo groups
Statistical Analysis 4: Comparison: Tramadol HCl/Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.0395, Wilcoxon (Mann-Whitney) — p-value for change from Baseline in general health at Day 29 was calculated for tramadol HCl/acetaminophen and placebo groups
Statistical Analysis 5: Comparison: Tramadol HCl/Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.0524, Wilcoxon (Mann-Whitney) — p-value for change from Baseline in vitality at Day 29 was calculated for tramadol HCl/acetaminophen and placebo groups
Statistical Analysis 6: Comparison: Tramadol HCl/Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.115, Wilcoxon (Mann-Whitney) — p-value for change from Baseline in social functioning at Day 29 was calculated using for tramadol HCl/acetaminophen and placebo groups
Statistical Analysis 7: Comparison: Tramadol HCl/Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.7788, Wilcoxon (Mann-Whitney) — p-value for change from Baseline in role emotional at Day 29 was calculated for tramadol HCl/acetaminophen and placebo groups
Statistical Analysis 8: Comparison: Tramadol HCl/Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.7776, Wilcoxon (Mann-Whitney) — p-value for change from Baseline in mental health at Day 29 was calculated for tramadol HCl/acetaminophen and placebo groups
Statistical Analysis 9: Comparison: Tramadol HCl/Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.0047, Wilcoxon (Mann-Whitney) — p-value for change from Baseline in Reptd. health transition at Day 29 was calculated for tramadol HCl/acetaminophen and placebo groups

5. Secondary Outcome: Change From Baseline in Oswestry Disability Index (ODI) Korean Version Score at Day 29
Description: The ODI Korean version was used to assess the participant's functionality. The ODI is a low back pain-specific, validated instrument that consists of questions related to limitations in performing specific activities of daily living and 1 question related to pain intensity. The ODI is a self-administered questionnaire consists of 10 sections. Each section consists of 6 statements ranked from 0 to 5 (0=good to 5=worse). Total score is the sum of score obtained in each section and ranges from 0 to 50. A higher score represents greater disability.
Time Frame: Baseline and Day 29
Population: FAS population included all participants who had received investigational product and had at least 1 data of measurement of primary efficacy endpoint.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Tramadol HCl/Acetaminophen | Placebo
Number analyzed (Participants) | 85 | 90
Unit on a scale
  Baseline | 39.626 (12.239) | 38.126 (13.518)
  Change at Day 29 (n=87,83) | 11.216 (11.856) | 7.178 (13.879)
Statistical Analysis 1: Comparison: Tramadol HCl/Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.0527, Wilcoxon (Mann-Whitney) — p-value for change from Baseline in ODI- Korean version at Day 29 was calculated for tramadol HCl/acetaminophen and placebo groups

6. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment on Investigational Product
Description: Global assessment on investigational product was done by investigator on how well the investigational product controlled chronic (lasting a long time) low back pain. Assessment was done by categories 'Very bad (-2)' 'Bad (-1)' 'Not changed (0) 'Good (1)' and 'Very good (2)'. Assessment better than "Good" was considered as pain improvement success. Percentage of participants with pain improvement success is reported here.
Time Frame: Day 29
Population: The FAS population included all the participants who had received investigational product and had at least 1 data of measurement of primary efficacy endpoint. Here 'N' signifies those participants who were evaluated for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tramadol HCl/Acetaminophen | Placebo
Number analyzed (Participants) | 80 | 83
Percentage of participants | 81.25 [72.70 to 89.80] | 69.88 [60.01 to 79.75]
Statistical Analysis 1: Comparison: Tramadol HCl/Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.0917, Chi-squared — p-value for investigator's global assessment on investigational product at Day 29 was calculated for tramadol HCl/acetaminophen and placebo groups

7. Secondary Outcome: Percentage of Participants With Participants' Global Assessment on Investigational Product
Description: Global assessment on investigational product was done by participants on how well the investigational product controlled chronic (lasting a long time) low back pain. Assessment was done by categories 'Very bad (-2)' 'Bad (-1)' 'Not changed (0) 'Good (1)' and 'Very good (2)'. Assessment better than "Good" was considered as pain improvement success. Percentage of participants with pain improvement success is reported here.
Time Frame: Day 29
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tramadol HCl/Acetaminophen | Placebo
Number analyzed (Participants) | 80 | 83
Percentage of participants | 76.25 [66.92 to 85.58] | 72.29 [62.66 to 81.92]
Statistical Analysis 1: Comparison: Tramadol HCl/Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.5632, Chi-squared — p-value for participant's global assessment on investigational product at Day 29 was calculated for tramadol HCl/acetaminophen and placebo groups

ADVERSE EVENTS:
Time Frame: Baseline up to Day 29
Arm/Group | Tramadol HCl/Acetaminophen | Placebo
Serious Adverse Events (participants affected / at risk) | 1/125 | 0/120
Other Adverse Events (participants affected / at risk) | 102/125 | 52/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tramadol HCl/Acetaminophen (N=125) | Placebo (N=120)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tramadol HCl/Acetaminophen (N=125) | Placebo (N=120)
Nasopharyngitis (Infections and infestations) | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 6 | 4
Headache (Nervous system disorders) | 11 | 6
Dizziness (Nervous system disorders) | 34 | 10
Somnolence (Nervous system disorders) | 18 | 4
Dysuria (Renal and urinary disorders) | 4 | 0
Dry mouth (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 45 | 12
Constipation (Gastrointestinal disorders) | 23 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 13 | 12
Thirst (General disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 6 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Cold sweating (Skin and subcutaneous tissue disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 21 | 5
Abdominal discomfort (Gastrointestinal disorders) | 0 | 4
Face oedema (General disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI cannot provide the any trial related information to external parties' without mutual agreement with the sponsor. This is valid even after the contract is canceled.